CLINICAL TRIAL: NCT04448587
Title: Sitagliptin for the Treatment of Grade 3-4 and Refractory Acute Graft-versus-host Disease
Acronym: GVHD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, moshe yeshurun, Head BMT Unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0368-20
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Graft Vs Host Disease
Keywords: SITAGLIPTIN
MeSH Terms: conditions — Graft vs Host Disease | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sitagliptin (Experimental)
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Sitagliptin 100mg — Oral sitagliptin will be commenced at a dose of 100 mg BID. The dose will be increased by 100 mg every three days up to a maximal dose of 300 mg BID. In the case of significant drug related side effects or drug intolerance, the last tolerated dose will be resumed. Patients responding well to lower doses of sitagliptin, will not be given higher doses of the drug. Sitagliptin will be provided as long as deemed effective by the treating physician up to three months.
  Other Names: JANUVIA

SUMMARY:
The prognosis of severe (grade 3-4) and steroid refractory acute graft-versus-host disease (GVHD) continues to be dismal. Sitagliptin given as GVHD-prophylaxis has recently been shown to reduce the incidence of acute GVHD to less than 10% with an excellent safety profile.

In this single center and single arm phase 2 study we aim to explore the safety and efficacy of sitagliptin in the treatment of severe and refractory acute GVHD.

Patient with new onset grade 3-4 acute GVHD will receive standard treatment consisting CNI and methylprednisolone 1-2 mg/kg/day or an equivalent dose of prednisone. Patients with refractory grade 2-4 acute GVHD will continue their current treatment; however methylprednisolone dose will be reduced to ≤ 1 mg/kg/day or an equivalent dose of prednisone.

Oral sitagliptin will be commenced at a dose of 100 mg BID. The dose will be increased by 100 mg every three days up to a maximal dose of 300 mg BID. In the case of significant drug related side effects or drug intolerance, the last tolerated dose will be resumed. Patients responding well to lower doses of sitagliptin, will not be given higher doses of the drug. Sitagliptin will be provided as long as deemed effective by the treating physician up to three months.

The primary end point will be the proportion of patients achieving complete remission(CR), very good partial response (VGPR) or partial response (PR) by day 28.

DETAILED DESCRIPTION:
The prognosis of severe (grade 3-4) and steroid refractory acute GVHD continues to be dismal. Sitagliptin given as GVHD-prophylaxis has recently been shown to reduce the incidence of acute GVHD to less than 10% with an excellent safety profile.

In this single center and single arm phase 2 study we aim to explore the safety and efficacy of sitagliptin in the treatment of severe and refractory acute GVHD.

Patient with new onset grade 3-4 acute GVHD will receive standard treatment consisting CNI and methylprednisolone 1-2 mg/kg/day or an equivalent dose of prednisone. Patients with refractory grade 2-4 acute GVHD will continue their current treatment; however methylprednisolone dose will be reduced to ≤ 1 mg/kg/day or an equivalent dose of prednisone.

Oral sitagliptin will be commenced at a dose of 100 mg BID. The dose will be increased by 100 mg every three days up to a maximal dose of 300 mg BID. In the case of significant drug related side effects or drug intolerance, the last tolerated dose will be resumed. Patients responding well to lower doses of sitagliptin, will not be given higher doses of the drug. Sitagliptin will be provided as long as deemed effective by the treating physician up to three months.

The primary end point will be the proportion of patients achieving CR, VGPR or PR by day 28. The secondary endpoints will be safety profile, proportion of patients achieving CR, VGPR or PR by day 56, 6-month duration of response (time from first response to GVHD progression or death), proportion of patients discontinuing immunosuppressive treatment by 3 and 6 months, proportion of patients developing chronic GVHD (limited and extensive) by 6 months, time to response, specific organ response, biomarker profile (ST2 and REG3a), Infection profile, OS at 6 months, GVHD free - disease free survival at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18-year old
* Grade 3-4 acute GVHD
* Refractory grade 2-4 acute GVHD
* Signed informed consent.
* Complete remission of the disease for which the patient was transplanted for.

Exclusion Criteria:

* Patients with diabetes mellitus requiring therapy with oral hypoglycemic medications or Insulin on top of sitagliptin.
* Serious hypersensitivity reaction to sitagliptin such as angioedema or anaphylaxis.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Response | day 28
  proportion of patients achieving complete remission (CR), very good partial response (VGPR) or partial response (PR) by day 28.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 3 months
  Incidence of treatment-emergent adverse events (safety and tolerability)
Response | day 56
  Proportion of patients achieving CR, VGPR or PR by day 56.
Response | 6 months
  GVHD free - disease free survival at 6 months
Biomarker profile | By days 0, 14, 28, 42, 56, 70, 100
  ST2 and REG3a blood levels

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No